CLINICAL TRIAL: NCT01677533
Title: Program for Research on the Outcomes of VA Education: Controlled Study of Panel Management and Microsystem Education Interventions to Improve Outcomes in Hypertension and Smoking Cessation
Brief Title: Program for Research on the Outcomes of VA Education
Acronym: PROVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA New York Harbor Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mark Schwartz, Primary Care Physician, VA New York Harbor Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EDU 08-428-2
Record Dates: First submitted 2012-08-28; First posted 2012-09-03 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Hypertension; Smoking Cessation
Keywords: Panel management; Clinical microsystems; Hypertension management; Smoking cessation; Continuing medical education; Quality improvement,; Population health
MeSH Terms: conditions — Hypertension; Smoking Cessation | interventions — Educational Status; Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PM-Data (Active Comparator): Team will receive data only.
  Interventions: Other: Data
- PM-Support (Experimental): Team will receive data and panel management support
  Interventions: Other: Data; Other: Panel Management Support
- PM-Education (Experimental): Team will receive data, panel management support, and educational interventions.
  Interventions: Other: Data; Other: Panel Management Support; Other: Education

INTERVENTIONS:
Other: Data — The microsystem teams of providers, nurses, and clerks will receive monthly reports of their performance measures, which will include process and outcome data for smoking cessation and blood pressure control for veterans in their panel. The reports will provide lists of individual patients in the panel with unmet goals on VA performance measures. They will receive written informational material describing principles and practices of panel management and evidence-based guidelines for hypertension management and smoking cessation.
Other: Panel Management Support — PMAs will meet regularly with the members of the microsystem team for one hour/week. The team will be asked to review progress on the health status of their patient panel and to plan strategies for improving their outcomes that the PMA will then implement. A PMA toolkit of panel management strategies will be established that will include guidelines for using VA databases to identify care gaps and reaching out to panel patients via phone and mail to intervene (e.g. reconnect patients to care with appointments, assess and enhance medication adherence, connect patients with VA services, motivational interviewing, and communication with the team about patient issues.
  Other Names: Panel management assistant
  Arms: PM-Education; PM-Support
Other: Education — The educational intervention will be administered throughout the duration of the study. Our initial educational focus will be on content (concepts of population health and panel management) and process (practice change methodology). Subsequent education will be process oriented, reviewing the changing system of care and discussing its functioning. Education will cover panel management strategies, microsystem theory and skills, and specific strategies regarding the management of hypertension and smoking cessation. It will include monthly seminars, reading materials, web-based modules, and skill building workshops, and PMA-conducted monthly academic detailing using panel data and feedback. After the first three months, academic detailing will only be implemented on an as-needed basis.
  Other Names: Educational Intervention
  Arms: PM-Education

SUMMARY:
The PROVE aims to test the efficacy of panel management support and educational intervention in VA Primary Care Clinical Microsystems. The study will test three increasingly intensive methods for implementing panel management strategies among health care providers in VA primary care clinics: providing only panel data, providing panel management support, and providing support plus clinical microsystem-enhancing education and training.It is hypothesized that the group receiving panel management and educational interventions will have better smoking cessation and hypertension outcomes than the group receiving only panel management assistance. It is further supposed that the later will have better smoking cessation and hypertension patient outcomes than the data-only group.

DETAILED DESCRIPTION:
Objective:

The specific aims for this study are: (1) to identify health professional educational and clinical microsystem determinants of outcomes for hypertension and smoking cessation in veterans. (2) to test the efficacy of three increasingly intensive methods for implementing panel management strategies among health care providers in VA primary care clinics: providing only panel data, providing panel management support, and providing support plus clinical microsystem-enhancing education and training.

Research design:

This project will consist of two phases. Phase I (one year) is the development of the necessary measurement and data infrastructure to assess health professional education, microsystem function, and clinical outcomes. In Phase 2 (two years) the study team will conduct a clinical demonstration project, comparing three interventions in a randomized controlled trial. Primary care teams will be randomly allocated to one of three arms: 1) panel management data, 2) panel management data and support, and 3) panel management data, support and education. The investigators will assess the impact of the implementation of panel management on primary patient outcomes in hypertension and smoking cessation (blood pressure and quit rates). The investigative team will also assess the impact of the implementation of panel management on secondary, intermediary, patient (patient activation, adherence, behavior change), provider (knowledge and attitudes, self-efficacy, job satisfaction) and microsystem outcomes (collective efficacy, teamwork, use of data, redesign of patient processes and provider roles/responsibilities, use of panel management strategies).

Methodology:

The study will utilize a multi-method, quasi-experimental design at VA NYHHS. Primary care is delivered through two teams at the Manhattan and five teams at the Brooklyn campuses. Patients, staff, nurses, and physicians are assigned to specific teams, thereby limiting contamination in this study.

ELIGIBILITY:
Inclusion Criteria:

* non-specialized primary care clinical microsystems

Exclusion Criteria:

* specialized clinical microsystems
* pilot clinical patient-aligned care teams

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5000 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2014-08-31 (Actual); Study Completion 2015-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Smoking Status | Baseline and 12 months
  clinical outcome
Change in Blood Pressure Reading | Baseline and 12 months
  clinical outcome

SECONDARY OUTCOMES:
Change in weight | Baseline and most recent at 12 months
Change in Patient Activation | 6 months and 12 months
  The Patient Activation Measure (PAM) is used to assess patients' self-reported knowledge, skill, and confidence in self-managing of health and chronic conditions
Change in Patient Perceptions of Quality of Care | 6 months and 12 months
Change in Provider Behavior change expertise | 6 months and 12 months
Change in Provider Self-efficacy with Panel Management Tasks | Baseline and 12 months
Change in Provider Job Satisfaction | Baseline and 12 months
Change in Microsystem function and collective efficacy | Baseline and 12 months
Change in Provider's assessments of training that they received in panel management and working within a PACT team | Baseline and 12 months
Change in Proportion of panel smokers offered smoking cessation resources by study arm | Baseline and 12 months
Change in Proportion of smokers on the panel received any cessation medications | Baseline and 12 months
  This information will be culled from the Vista Smoking Database

OTHER OUTCOMES:
Change in Health care usage | Baseline and 12 months
  Number of primary care visits, mental health visits, emergency room/urgent care visits and the number of VA hospitalizations
Change in Patient-level costs | Baseline and 12 months
  Outpatient primary care visits, mental health visits, pharmacy and hospitalizations from the VA Decision Support System

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Schwartz, Principal Investigator — VA New York Harbor Healthcare System; Scott Sherman, M.D., M.P.H., Principal Investigator — VA New York Harbor Healthcare System; Colleen Gillespie, PhD, Study Director — NYU Langone Health; Anne Dembitzer, M.D., Study Director — VA New York Harbor Healthcare System
Locations (2):
- United States (2):
  - VA NYHHS Brooklyn Campus, Brooklyn, New York
  - VA NYHHS Manhattan Campus, New York, New York

REFERENCES:
- [Derived] Savarimuthu SM, Jensen AE, Schoenthaler A, Dembitzer A, Tenner C, Gillespie C, Schwartz MD, Sherman SE. Developing a toolkit for panel management: improving hypertension and smoking cessation outcomes in primary care at the VA. BMC Fam Pract. 2013 Nov 21;14:176. doi: 10.1186/1471-2296-14-176. PMID 24261337